CLINICAL TRIAL: NCT06448195
Title: Growth Hormone Replacement Therapy on Metabolic Effects in Patients With Fatty Liver Caused by Growth Hormone Deficiency After Pituitary GH Adenoma Surgery: A Monocentric, Prospective, Randomized, Parallel-controlled Clinical Study.
Brief Title: Effects of Growth Hormone Therapy on Metabolic Function in Fatty Liver Post-Pituitary Adenoma Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-071R2
Record Dates: First submitted 2024-05-28; First posted 2024-06-07 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Growth Hormone Treatment
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth hormone treatment group (Experimental): A total of 20 patients with liver fat content greater than 11% determined by proton magnetic resonance spectroscopy (1H MRS) method were recruited six months to two years after operation of pituitary adenoma, and underwent growth hormone replacement therapy, the total course of treatment was 6 months, and finally the liver fat content was determined
  Interventions: Drug: Polyethylene Glycol Somatropin (rDNA origin) Injection
- Lifestyle intervention control group (No Intervention): A total of 20 patients with liver fat content greater than 11% determined by proton magnetic resonance spectroscopy (1H MRS) method were recruited six months to two years after operation of pituitary adenoma. The patients were treated as the control group and underwent lifestyle intervention. Finally, the liver fat content was determined

INTERVENTIONS:
Drug: Polyethylene Glycol Somatropin (rDNA origin) Injection — Specification: 54IU/9.0mg/1.0ml/ bottle Dosage form: injection; Dose: 1mg/ week. Subcutaneous injection (upper arm, thigh or abdomen periumbilical) for a total course of 6 months, a total of 3 bottles per patient
  Other Names: Growth hormone replacement therapy
  Arms: Growth hormone treatment group

SUMMARY:
Growth Hormone (GH) is essential for maintaining fat, muscle, bone, and energy balance. Adult Growth Hormone Deficiency (GHD) affects about 0.3% of adults. GHD, common post-pituitary tumor surgery or radiotherapy, disrupts lipid metabolism, increasing triglycerides and low-density lipoprotein cholesterol while decreasing high-density lipoprotein cholesterol. This is especially severe in GH adenoma patients, whose lipid metabolism issues worsen post-surgery, increasing the risk of atherosclerosis. Fat accumulates in the liver first, making liver fat content a key early indicator of metabolic disorders, which can lead to diabetes and atherosclerosis. Early intervention is crucial as liver fat deposition in Nonalcoholic Fatty Liver Disease (NAFLD) is reversible.

Recombinant human growth hormone can treat GHD-related lipid metabolism disorders, but research on its effects on liver fat in post-surgery GH adenoma patients is limited. The investigators plan to treat these patients with 1 mg/week of recombinant human growth hormone for 24 weeks, aiming to normalize insulin-like growth factor-1 levels. Liver fat content changes will be measured using proton magnetic resonance spectroscopy (1H MRS) and Fibroscan. Changes in weight, BMI, waist circumference, fasting blood glucose, blood lipids, and other metabolic factors will also be evaluated to assess treatment efficacy and safety.

Zhongshan Hospital, affiliated with Fudan University, performs over 300 pituitary tumor surgeries annually, including 100 GH adenoma cases. The hospital has extensive experience and can enroll 40 patients. The Endocrinology Department excels in evaluating lipid metabolism disorders in NAFLD using non-invasive methods. As a major hospital in Shanghai, it has ample patients to meet study requirements. Detailed exit criteria and rescue plans have been established to address potential adverse events during the study.

DETAILED DESCRIPTION:
Growth Hormone (GH) is an important hormone secreted by the pituitary gland and is essential for maintaining normal fat, muscle, bone content, and energy balance in the body. The prevalence of adult Growth Hormone Deficiency (GHD) is approximately 0.3% in adults. When human growth hormone is deficient, lipid metabolism is most prone to disorder. The study found that blood triglyceride and low-density lipoprotein cholesterol levels increased in GHD patients, and blood high-density lipoprotein cholesterol levels decreased. GHD is most common in patients with pituitary tumor after surgery or radiotherapy, especially in patients with GH adenoma after surgery. The lipid metabolism disorder is the most serious among all GHD patients because the excessive growth hormone before surgery has caused a state of severe lipid metabolism disorder, and after surgery, patients are directly converted to a state of growth hormone deficiency, exacerbating the lipid metabolism disorder. This disorder will progress from poor to worse, and long-term follow-up shows a higher likelihood of developing secondary atherosclerotic diseases post-surgery.

Current studies have shown that when abnormal lipid metabolism occurs in GHD patients, fat will first accumulate in the liver. Therefore, compared with changes in blood lipid metabolism indexes and body components, changes in liver fat content can detect abnormal lipid metabolism earlier. Liver fat deposition, as the initiating factor of systemic metabolic disorders, is involved in the occurrence and development of diabetes and atherosclerotic diseases. Currently, it is considered that the fat deposition in Nonalcoholic Fatty Liver Disease (NAFLD) is reversible. Therefore, it is particularly urgent to conduct very early intervention for GHD patients with pituitary GH adenoma after operation to block the occurrence of subsequent metabolic adverse events.

It has been reported that recombinant human growth hormone can be used in the treatment of abnormal lipid metabolism due to GHD, but at present, there is a lack of relevant studies on recombinant human growth hormone in the treatment of abnormal lipid metabolism in patients with pituitary GH adenoma after surgery, especially the study on the change of liver fat content. The investigators intend to apply a recombinant human growth hormone dose of 1 mg/week (6 IU is 1 mg) to GH adenoma patients with GHD and NAFLD after GH adenoma surgery, aiming to increase the insulin-like growth factor-1 of patients to the median of the normal level of peers, with a treatment duration of 24 weeks. After treatment, changes in liver fat content at baseline and 24 weeks after intervention will be measured by proton magnetic resonance spectroscopy (1H MRS) and Fibroscan liver stiffness. The changes in metabolic parameters (body weight, body mass index (BMI), waist circumference, fasting blood glucose, blood lipids, high iron content, and other metabolic-related inflammatory factors) before and after recombinant human growth hormone treatment will be evaluated.

This study aims to evaluate the efficacy and safety of recombinant human growth hormone in the treatment of GHD-induced NAFLD patients with abnormal lipid metabolism after GH adenoma surgery and propose a suitable treatment method for people with abnormal lipid metabolism due to GHD after GH adenoma surgery, providing a direct basis for establishing a standardized clinical treatment path in the next step.

The Department of Neurosurgery of Zhongshan Hospital Affiliated to Fudan University carries out more than 300 cases of various types of pituitary tumors every year, including more than 100 cases of pituitary GH adenoma. It has developed a multidisciplinary joint clinic for pituitary tumors earlier in China and has rich experience in the diagnosis and treatment of pituitary tumors, meeting the needs of 40 enrolled cases. The Department of Endocrinology has been committed to the evaluation of lipid metabolism disorders in nonalcoholic fatty liver for a long time. Currently, ultrasound and imaging are proficient in non-invasive methods of determining liver fat, such as MRS liver stiffness test. As a large Class III hospital in Shanghai, with a wealth of pituitary tumor patients, it can meet the enrollment requirements of subjects, and the endocrinology department can complete the assessment of lipid metabolism disorder. Detailed exit criteria and rescue plans have been jointly developed. Adverse events that may occur during the study were defined and addressed in detail.

ELIGIBILITY:
Inclusion Criteria:

* Have fully understood the informed consent and signed the informed consent;
* Age: 18-60 years old;
* Patients diagnosed with adult growth hormone deficiency (AGHD) (GH stimulation test: GH peak ≤5ug/l or organic hypothalamic-pituitary disease ≥3 pituitary hormone deficiency with IGF-1 < -2SD)
* Patients with pituitary growth hormone adenoma proved pathologically after surgery
* Anterior pituitary hormone supplementation (except growth hormone)
* The liver fat content was more than 11% after six months to two years of operation by proton magnetic resonance spectroscopy (1H MRS).
* Those who have not taken lipid-regulating drugs (statins, Bates);
* Blood pressure <150/95mmHg, did not take any antihypertensive drugs;

Exclusion Criteria:

* Have any of the following liver disease history: chronic hepatitis, cirrhosis, liver cancer, autoimmune liver disease, alcoholic liver disease, hereditary liver disease
* Significant abnormal liver function: ALT or AST≥ 2 times the upper limit of normal; HBsAg (+), and/or HCV-Ab (+);
* Patients with serum creatinine value ≥1.5mg/dL (133umol/L);
* Patients with severe heart disease (patients with a history of myocardial infarction and heart failure and/or severe arrhythmia);
* Patients with severe infection, other operations within 6 months, or severe trauma;
* Alcohol consumption (alcohol): male ≥140g/week; Female ≥70g/week;
* Poorly controlled diabetic patients: HbA1c >9.5% within three months; Or use hypoglycemic drugs that may affect liver histopathology, including pioglitazone, GLP-1, and DP-4 inhibitors;
* Patients with allergy or intolerance to the same drug used in the trial;
* In the next 1 year, there are pregnancy plans or breastfeeding patients or patients with mental disorders;
* Patients who have participated in other clinical trials within 24 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the percentage of liver fat | up to 6 months
  To evaluate the effect of recombinant growth hormone replacement therapy on hepatic fat content in NAFLD patients with GHD after pituitary GH adenoma surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xie, Study Director — Fudan University
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China